CLINICAL TRIAL: NCT03982472
Title: Shoulder Transcutaneous Electric Nerve Stimulation Decelerates Heart Rhythm of Subjects Via Potentiating Vagal Tone
Brief Title: TENS Impact Heart Rate Via Vagus Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Tzer-Bin Lin, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TENS-HR
Record Dates: First submitted 2019-06-10; First posted 2019-06-11 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Transcutaneous Electric Nerve Stimulation; Heart Rate
Keywords: heart rate; TENS; vagus nerve
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Difference of group was compared between groups
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TENS right side (Experimental): TENS stimulation at the right side
  Interventions: Other: transcutaneous electric stimulation
- TENS left side (Experimental): TENS stimulation at the left side
  Interventions: Other: transcutaneous electric stimulation
- sham stimulation (No Intervention): Sham stimulation

INTERVENTIONS:
Other: transcutaneous electric stimulation — transcutaneous current with an amplitude around ten to hundred milliampere was applied topically to subjects
  Arms: TENS left side; TENS right side

SUMMARY:
Transcutaneous electric nerve stimulation (TENS) is widely used for the treatment of adhesive capsulitis, nevertheless, its potential impact on heart physiology has not been well established.

The investigator explored if TENS at shoulder region affect heart rhythm and the machinery involved.

Subjects were stratified into groups received sham stimulation (TENS-S) and TENS on either the right (TENS-R) or left (TENS-L) shoulder. A built-in waveform for treating adhesive capsulitis with a maximal tolerable intensity below the pain threshold was applied to subjects form a commercial TENS equipment for 5 min. The electrocardiogram (ECG) and heart rate (HR) were continuously recorded and the ECG was off-line transferred into power spectrum for analysis.

DETAILED DESCRIPTION:
Study design This study complied with the Declaration of Helsinki, and all protocols were approved by the ethics committee of Taoyuan General Hospital, Ministry of Health and Welfare, Taoyuan, Taiwan. All the participants gave written informed consent before experiments. 32 subjects (20-51 years old) were included in the statistical analysis. Participants were eligible if they have cardiovascular illnesses, major mental conditions, or severe inflammation. Participants were allocated to groups that received sham stimulation (TENS-S) and TENS on the right and left shoulder (TENS-R and TENS-L, respectively).

ECG and HR recordings Using a monitor lead, electrocardiogram (ECG) was recorded through electrodes connected to a recording system with a sampling rate of 5,000 samples/sec. The ECG and the HR calculated by a built-in rate meter were continuously recorded and displayed on a monitor. For TENS caused marked artifacts in ECG tracings, HR derived from ECG were confirmed off-line by manual examination.

TENS stimulation To mimicking clinical scenarios, a commercial TENS equipment was used throughout this study. A built-in waveform recommended for treating capsulitis in the user's manual was used for stimulation (triple pulses with 1 ms pulse durations separated by a 1 ms intervals were ramps up and down between 2 to 10 Hz within 20 sec for 3 min and then ramps up from 10 to 200 Hz within 20 sec and kept at 200 Hz for 2 min; supplementary data 1). The current intensity was adjusted to the maximal tolerance level below the pain threshold. A pair of stimulating electrode was placed in the front of the should at the level of the sternal notch at about 2 finger-width from the mid-clavicle line, and a pair of dispersive electrode was placed at the back of shoulder opposite to the stimulating electrodes. Participants kept a stationary supine position and was asked to refrain from moving during recording. Before the stimulation, there was an equilibrium period for at least 10 min, and then the recording started. TENS was turned on for 5 min at 5 min after the baseline recording, and the recording continued until 10 min after the offset of stimulation. Parameters of the sham stimulation was identical to TENS stimulation on the right shoulder excepting the equipment was left un-powered.

ELIGIBILITY:
Inclusion Criteria:

healthy adult

Exclusion Criteria:

hypertension diabetes heart diseases neurological diseases othe medical problem

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-22 (Actual); Primary Completion 2018-07-21 (Actual); Study Completion 2018-07-21 (Actual)

PRIMARY OUTCOMES:
heart rate | 5 min
  TENS stimulation modified HR

CONTACTS AND LOCATIONS:
Overall Officials: Tzer-Bin Lin, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
After our results have been published

REFERENCES:
- [Background] Badran BW, Mithoefer OJ, Summer CE, LaBate NT, Glusman CE, Badran AW, DeVries WH, Summers PM, Austelle CW, McTeague LM, Borckardt JJ, George MS. Short trains of transcutaneous auricular vagus nerve stimulation (taVNS) have parameter-specific effects on heart rate. Brain Stimul. 2018 Jul-Aug;11(4):699-708. doi: 10.1016/j.brs.2018.04.004. Epub 2018 Apr 6. PMID 29716843
- [Background] Brock C, Brock B, Aziz Q, Moller HJ, Pfeiffer Jensen M, Drewes AM, Farmer AD. Transcutaneous cervical vagal nerve stimulation modulates cardiac vagal tone and tumor necrosis factor-alpha. Neurogastroenterol Motil. 2017 May;29(5). doi: 10.1111/nmo.12999. Epub 2016 Dec 12. PMID 27957782
- [Background] Connor DE Jr, Nixon M, Nanda A, Guthikonda B. Vagal nerve stimulation for the treatment of medically refractory epilepsy: a review of the current literature. Neurosurg Focus. 2012 Mar;32(3):E12. doi: 10.3171/2011.12.FOCUS11328. PMID 22380853
- [Derived] Hsieh CM, Lin WC, Peng HY, Chen HC, Ho YC, Li CJ, Wu XG, Chung JY, Lee SD, Lin TB. Shoulder transcutaneous electric nerve stimulation decreases heart rate via potentiating vagal tone. Sci Rep. 2021 Sep 27;11(1):19168. doi: 10.1038/s41598-021-98690-6. PMID 34580404